CLINICAL TRIAL: NCT07270991
Title: Randomized Phase III Trial to Compare Trifluridine/Tipiracil + Fruquintinib Versus Trifluridine/Tipiracil Alone for Metastatic Oeso-gastric Adenocarcinoma
Brief Title: Trifluridine/Tipiracil + Fruquintinib Versus Trifluridine/Tipiracil Alone for Metastatic Oeso-gastric Adenocarcinoma
Acronym: FRUQUITAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGIC06-PRODIGE114-FRUQUITAS; 2025-522395-92-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Oesogastric Adenocarcinoma
Keywords: Cancer; Fruquintinib; oeso-gastric; third line
MeSH Terms: conditions — Neoplasms | interventions — trifluridine tipiracil drug combination; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (control arm): trifluridine/tipiracil (Active Comparator): Cycle of 28 days 35 mg/m2 by mouth twice daily on Days 1 to 5, 2 days of rest and 35 mg/m2 by mouth twice daily on days 8 to 12
  Interventions: Drug: trifluridine/tipiracil
- Arm B (experimental arm): trifluridine/tipiracil + fruquintinib (Experimental): Cycle of 28 days
  For trifluridine/tipiracil: 35 mg/m2 by mouth twice daily on Day 1 to 5, 2 days of rest and 35 mg/m2 by mouth twice daily on days 8 to 12
  For fruquintinib: 5 mg by mouth once daily Day 1 to Day 21 (3 weeks) Treatment will be repeated every 4 weeks until radiological disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: trifluridine/tipiracil; Drug: fruquintinib

INTERVENTIONS:
Drug: trifluridine/tipiracil — Cycle of 28 days 35 mg/m2 by mouth twice daily on Days 1 to 5, 2 days of rest and 35 mg/m2 by mouth twice daily on days 8 to 12 Treatment will be repeated every 4 weeks until radiological disease progression, unacceptable toxicity or patient's refusal.
Drug: fruquintinib — For fruquintinib: 5 mg by mouth once daily Day 1 to Day 21 (3 weeks) Treatment will be repeated every 4 weeks until radiological disease progression, unacceptable toxicity or patient's refusal.
  Arms: Arm B (experimental arm): trifluridine/tipiracil + fruquintinib

SUMMARY:
Advanced cancer of the stomach and the gastro-esophageal junction (G/GEJ) remains a very serious disease. Today, only about 10-15% of patients are alive after 5 years. Treatments mainly aim to control symptoms, extend life, and maintain quality of life.

First treatments usually combine two chemotherapies, but recent years have brought real progress. Immunotherapy - drugs that "unlock" the immune system - has shown clear benefits. For patients whose tumors have certain markers (like PD-L1), combining drugs such as nivolumab or pembrolizumab with chemotherapy can help patients live longer. Another breakthrough is zolbetuximab, a targeted therapy that attacks a protein (Claudin 18.2) found on many gastric cancers, also improving survival.

When cancer grows despite these therapies, second-line treatments are used. The most common is chemotherapy with paclitaxel + ramucirumab, which blocks the tumor's blood supply. These drugs extend survival, but usually only by a few months.

For patients who need a third option, the oral drug trifluridine/tipiracil (TAS-102) can provide extra time, though benefits remain limited. That's why researchers are now exploring combinations. Since stomach tumors rely on forming new blood vessels, combining trifluridine/tipiracil with anti-angiogenic drugs - medicines that cut off the tumor's blood supply - looks promising.

One of the most exciting of these drugs is fruquintinib, already proven effective in colorectal cancer. A new international trial, FRUQUITAS (ENGIC 06/PRODIGE 114), is now testing whether adding fruquintinib to trifluridine/tipiracil can improve survival for patients with advanced stomach or gastro-esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (patients enrolled gender independently).
2. Histologically proven metastatic adenocarcinoma of the stomach or the esophagogastric junction (GEJ) or esophagus.
3. Prior treatment by two or three lines of treatment for metastatic setting (patients who received adjuvant therapy and developed metastatic disease within 6 months of completing treatment should be considered as having failed first-line therapy for metastatic disease).
4. Prior treatment (progression or intolerance) with platinum salts (oxaliplatin or cisplatin), fluoropyrimidine and irinotecan and/or taxane (+/- anti-HER2 agents +/- immune checkpoint inhibitors +/- ramucirumab +/- anti-claudin 18.2).
5. Measurable or non-measurable lesions. (Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
6. World Health Organisation (WHO) performance status 0-1.
7. Adequate organ function: ANC ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dL, platelets ≥ 100 G/L, AST/ALT ≤ 3 x ULN (≤ 5 x ULN in case of liver metastase(s)), total bilirubin ≤ 1.5 x ULN, creatinine clearance > 30 mL/min (CKD EPI).
8. Adequate coagulation tests (INR and activated partial thromboplastin time (APTT) ≤1.5 × ULN) unless the patient is receiving anticoagulant therapy.
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.
10. Man and woman of childbearing potential agrees to use two methods (one for the patient and one for the partner) of medically acceptable forms of contraception (use contraceptive methods that result in a failure rate of <1% per year) during the study and for 6 months after the last treatment intake.
11. Patient is able to understand, sign, and date the written informed consent form at the screening visit prior to any protocol-specific procedures performed.
12. Available tumor block (surgical specimens of primary tumor and if not available tumor biopsies).
13. Patient willing to participate to biological studies.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study - unless it is an observational study or during the follow-up for survival status update only of an interventional study.
2. Administration of the last dose of anticancer therapy and palliative radiotherapy ≤ 2 weeks prior to the first dose of study drug.
3. Current or prior bowel obstruction within 28 days before the first dose of study drugs.
4. Any unresolved clinical significant toxicity NCI CTCAE v5.0 ≥ grade 2 from previous anticancer therapy (except neuropathy).
5. More than 3 prior lines of treatment.
6. Major surgical procedure (e.g. exploratory laparoscopy is not considered as a major surgical procedure) within 2 weeks prior to the first dose of treatment.
7. History of leptomeningeal carcinomatosis or symptomatic or untreated brain metastase(s). Patients whose brain metastase(s) have been treated may participate if any neurologic symptoms that developed as a result of the brain metastases are resolved or stable.
8. Severe cardiac disorders (including but not limited to acute myocardial infarction, stroke, unstable angina, NYHA class III/IV heart failure, or LVEF<50%) within 6 months.
9. Severe liver dysfunction (cirrhosis Child Pugh B or C).
10. Gastric or duodenal active ulcer.
11. Thromboembolic events (including deep vein thrombosis and pulmonary embolism) in the past 6 months
12. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled hypertension (defined as systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg despite optimal medical management), interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea,
13. psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. Patients with urine protein test 2+ or more and 24 hours urine protein≥1.0g/24h.
15. Known positive test for HIV, active hepatitis B or hepatitis C, active tuberculosis.
16. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients (excipients with known effects and potential risk of allergies : tartrazine (E102) ,sunset yellow FCF (E110), Lactose monohydrate).
17. Prior treatment with trifluridine/tipiracil and/or fruquintinib and/or regorafenib and/or any anti-VEGFR tyrosine kinase inhibitor.
18. Active infection requiring intravenous antibiotics at the time of Day 1 of Cycle 1.
19. Other malignancy within 3 years prior to study enrolment, except for localized cancer in situ, basal or squamous cell skin cancer or other localized tumor with complete resection.
20. Treatment with powerful CYP 450 inducers (no contraindication for inhibitors).
21. Pregnant or breastfeeding female patient.
22. Congenital galactosemia, total lactase deficiency (lactose intolerance) or glucose-galactose malabsorption syndrome.
23. Patients with clinically significant bleeding within the past 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 18 months after randomization
  The primary endpoint is the Overall survival (OS) and is defined as the time between the date of randomization and the date of death caused by any reason or the date of last news if the patient is alive.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up 18 months after randomization
  Progression-free survival (PFS) is defined as the time between date of randomization and the date of first radiological progression according to RECIST 1.1 or death (whichever occurs first). Patients alive without progression will be censored to the date of last radiologic assessment.

CONTACTS AND LOCATIONS:
Locations (64):
- France (56):
  - Centre Hospitalier, Aurillac
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier, Bayeux
  - Bayonne- Clinique Belharra, Bayonne
  - Centre Hospitalier Côte Basque, Bayonne
  - ICONE, Bezannes
  - BORDEAUX-Institut Bergonié, Bordeaux
  - Clinique Tivoli, Bordeaux
  - C.H.U. de Brest, Brest
  - Cac - François Baclesse, Caen
  - CHU Côte de Nacre, Caen
  - Ch - Jean Rougier, Cahors
  - Centre Hospitalier, Cholet
  - Saint Côme, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - Centre Leonard de Vinci, Dechy
  - Institut de cancérologie de Bourgogne GRReCC, Dijon
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Hôpital Franco-Britannique, Levallois-Perret
  - CHU Dupuytren, Limoges
  - Groupement Hospitalier Bretagne Sud, Lorient
  - Hôpital Prive Jean Mermoz, Lyon
  - Chu - Hôpital La Timone, Marseille
  - CAC Paoli Calmettes, Marseille
  - Confluent Sas, Nantes
  - CAC Antoine Lacassagne, Nice
  - Gh Nord Essone, Orsay
  - Privé - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Chu - Aphp - Hôpital Saint Louis, Paris
  - Chu - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Cochin (APHP), Paris
  - Centre Hospitalier, Pau
  - Centre Hospitalier Saint Jean, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chu - Centre Hospitalier Universitaire de Poitiers - La Miletrie, Poitiers
  - Clinique de La Croix du Sud, Quint-Fonsegrives
  - Chu - Centre Hospitalier Universitaire Robert Debre, Reims
  - CAC Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Polyclinique, Rillieux-la-Pape
  - CHU - Charles Nicolle, Rouen
  - Clinique Mathilde, Rouen
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Ch Memorial France Etats Unis, Saint-Lô
  - Hia Begin, Saint-Mandé
  - Clinique Mutualiste de L'Estuaire, Saint-Nazaire
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Center Hospitalier de Sens, Sens
  - Groupe Hospitalier Rance Emeraude, St-Malo
  - CAC - Paul Strauss, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Hôpital FOCH, Suresnes
  - Hia Sainte Anne, Toulon
  - CHRU de Tours - Hopital Trousseau, Tours
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
  - Ch Nord Ouest, Villefranche-sur-Saône
- Germany (8):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Haematologisch Onkologische Praxis Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Uniklinikum Leipzig, Leipzig
  - Klinikum Rechts Der Isar Der Technischen Universitat Munchen, München
  - Rostock University Medical Center, Rostock

IPD SHARING:
Plan to Share IPD: No